CLINICAL TRIAL: NCT02003794
Title: Randomized Controlled Study of the Effectiveness of IV Fluid Infusion in Patients With Acute Ischemic Stroke (IVIS)
Acronym: IVIS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: More progressive stroke in one arm
Sponsor: Chulalongkorn University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Principal Investigator, Nijasri C Suwanwela, Division of Neurology, Department of Medicine, Faculty of Medicine, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IVIS 001
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Ischemic Stroke
Keywords: acute ischemic stroke; intravenous fluid; ้hydration
MeSH Terms: conditions — Ischemic Stroke | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV Fluid (Experimental): 0.9% NaCl solution infusion: 100 ml/hr for three days.
  Interventions: Drug: 0.9% NaCl solution
- No IV Fluid (No Intervention): Not receive any intravenous fluid but can consume oral fluid normally for three days.

INTERVENTIONS:
Drug: 0.9% NaCl solution — 0.9% NaCl solution intravenous infusion: 100 ml/hr for three days.
  Other Names: Normal saline
  Arms: IV Fluid

SUMMARY:
To study the result of intravenous fluid in patients with acute ischemic stroke within 72 hours.

DETAILED DESCRIPTION:
This study aims to find the effect of early IV fluid administration to patients with acute ischemic stroke on the neurological outcome and to determine the side effects of intravenous fluids. Due to its cost effectiveness and wide accessibility, the possible application or use of IV fluid infusion as first line treatment can aide in the treatment of more acute ischemic stroke patients worldwide. This novel information will aide physicians with more comprehensive understanding of the efficacy of utilizing IV fluid in future treatment plans for patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18-80 years
2. NIHSS ≥ 1
3. Diagnosis of acute ischemic stroke within 72 hours from stroke onset
4. Enrollment into the study within 24 hours after hospital arrival
5. Urine specific gravity level < 1.030
6. Patient consent

Exclusion Criteria:

1. Patients receiving > 40 ml/hr IV fluid infusion over 3 hours
2. Acute ischemic stroke caused cardiogenic embolism
3. Urine specific gravity ≥ 1.030
4. Large cerebral infarction area

   1. Infarction > 1/3 of middle cerebral artery area
   2. Infarction > 1/2 of cerebellar hemisphere
5. NHISS ≥ 18
6. Previous or current episode of atrial fibrillation
7. Previous or current episode congestive heart failure
8. Previous echocardiogram with ejection fraction < 40%
9. Previous or current episode of dilated cardiomyopathy
10. Abnormal renal function GFR ≤ 60% or serum creatinine ≥ 2
11. Modified Rankin scale before acute ischemic stroke ≥ 2
12. Patients receiving intravenous thrombolysis
13. NPO with need for IV fluid
14. IV fluid infusion needed from any other causes
15. Patients with poor prognosis with life expectancy < 90 days
16. Patients involved in other ongoing clinical studies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
NIHSS ≤ 4 | day 7 after treatment or on the day of discharge
  Patients with good outcome by NIHSS ≤ 4 at day 7 after treatment or on the day of discharge, which ever comes first.

SECONDARY OUTCOMES:
mRS ≤ 1 | day 7 after treatment or on the day of discharge
  Patients with mRS ≤ 1 at day 7 after treatment or on the day of discharge, which ever comes first.
mRS ≤ 4 | at day 90
  Patients with mRS ≤ 4 at day 90
mRS ≤ 1 | at day 90
  Patients with mRS ≤ 1 at day 90
change of serum osmolarity | at day 3 after treatment
  Percentage of change of serum osmolarity at day 3 after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nijasri C Suwanwela, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn University, Bangkok, Bangkok, Thailand